CLINICAL TRIAL: NCT02825134
Title: Nordic Aortic Valve Intervention Trial 2 - A Randomized Multicenter Comparison of Transcatheter Versus Surgical Aortic Valve Replacement in Younger Low Surgical Risk Patients With Severe Aortic Stenosis
Brief Title: Comparison of TAVR With SAVR in Younger Low Surgical Risk Patients With Severe Aortic Stenosis
Acronym: NOTION-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ole De Backer (Other)
Collaborators: Symetis SA (Industry); Boston Scientific Corporation (Industry); Abbott (Industry); Edwards Lifesciences (Industry)
Responsible Party: Sponsor-Investigator, Ole De Backer, MD, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-15019580
Record Dates: First submitted 2016-06-29; First posted 2016-07-07 (Estimated); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Aortic Valve Stenosis; Cardiovascular Diseases; Heart Diseases; Heart Valve Diseases; Ventricular Outflow Obstruction
Keywords: heart valve disease; valvular bioprosthesis; aortic valve replacement; Randomized clinical trial
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases; Heart Diseases; Heart Valve Diseases; Ventricular Outflow Obstruction | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcatheter aortic valve replacement (Experimental): Transcatheter aortic valve replacement
  Interventions: Device: Transcatheter aortic valve replacement
- Surgical aortic valve replacement (Active Comparator): Surgical aortic valve replacement
  Interventions: Device: Surgical aortic valve replacement

INTERVENTIONS:
Device: Transcatheter aortic valve replacement — Retrograde transfemoral transcatheter aortic valve replacement with any CE mark approved aortic bioprosthesis with or without concomitant percutaneous coronary intervention.
  Other Names: Transcatheter aortic valve implantation; TAVR; TAVI
  Arms: Transcatheter aortic valve replacement
Device: Surgical aortic valve replacement — Conventional surgical aortic valve replacement with a bioprosthesis using normothermic cardiopulmonary bypass and cold blood cardioplegia cardiac arrest with or without concomitant coronary artery bypass graft surgery.
  Other Names: SAVR
  Arms: Surgical aortic valve replacement

SUMMARY:
A randomized clinical trial investigating transcatheter (TAVR) versus surgical (SAVR) aortic valve replacement in patients 75 years of age or younger suffering from severe aortic valve stenosis.

Study hypothesis: The clinical outcome (death of any cause, stroke and rehospitalization (related to the procedure, valve or heart failure)) obtained within one year after TAVR is non-inferior to SAVR.

DETAILED DESCRIPTION:
BACKGROUND: Acquired aortic valve stenosis (AS) is the most common heart valve disease in the Western World with a prevalence of 2-7% at the age of >65 years. If untreated, it may lead to heart failure and death. Surgical aortic valve replacement (SAVR) until recent years has been the definitive treatment for patients with severe symptomatic AS. A less invasive transcatheter aortic valve replacement (TAVR) has been developed and has been a treatment of choice mostly for elderly high risk or inoperable patients. As TAVR technology is continuously evolving and improving, it may be anticipated that it will become a valuable alternative - and even the preferred choice of treatment - for younger, low-risk patients with severe aortic valve stenosis in the near future. However, to date, there is no clinical evidence that supports this hypothesis.

AIM: The purpose of the study is to compare TAVR and SAVR with regard to the intra- and post-procedural morbidity and mortality rate, hospitalization length, functional capacity, quality of life, and valvular prosthesis function in younger, low risk patients with severe bicuspid or tricuspid AS, scheduled for aortic valve replacement.

POPULATION: Younger low risk patients with severe aortic valve stenosis, which are scheduled for aortic valve replacement using a bioprosthesis. Subjects fulfilling the inclusion criteria, not having any exclusion criteria, and consenting to the trial will be randomized 1:1 to TAVR or SAVR with 186 patients in each group.

DESIGN: The study is a randomized clinical multicenter trial. Central randomization with variable block size and stratification by gender and coronary comorbidity will be used. An independent event committee blinded to treatment allocation will adjudicate safety endpoints.

INTERVENTIONS:

TAVR: Any CE-Mark approved transcatheter aortic bioprosthesis may be used in the study, and the choice is at the discretion of the local TAVR team. The transfemoral TAVR procedure may be performed under general anaesthesia, local anaesthesia/conscious sedation, or local anesthesia. Percutaneous coronary intervention (PCI) can be performed up to 30 days prior to TAVR or as a hybrid procedure.

SAVR: The surgical SAVR technique follows standard protocol of the local department of cardio-thoracic surgery. The operation is performed under general anesthesia, which follows standard protocol of the department of anesthesiology. A commercial available surgical aortic bioprosthesis at the surgeons discretion will be implanted. Concomitant coronary artery bypass graft (CABG) surgery may be performed.

END POINTS: The primary endpoint is the composite rate of death of any cause, stroke and rehospitalization (related to the procedure, valve or heart failure) within one year after the procedure. Secondary endpoints are listed below. Follow-up will be performed after 1 and 12 months and yearly thereafter for a minimum of 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 75 years or younger.
* Severe calcific AS (Valve area <1cm2 (or <0.6 cm2/m2) AND one of the two following criteria: mean gradient >40mmHg or peak jet velocity >4.0m/s, OR in presence of low flow, low gradient with reduced or normal LVEF<50%, a dobutamine stress echo should verify true severe AS rather than pseudo-AS
* Symptomatic with angina pectoris, dyspnea or exercise-induced syncope or near syncope OR asymptomatic with abnormal exercise test showing symptoms on exercise clearly related to AS or systolic LV dysfunction (LVEF <50%) not due to another cause.
* Anticipated usage of biological aortic valve prosthesis.
* Low risk for conventional surgery (STS Score <4%).
* Suitable for both SAVR and transfemoral TAVR.
* Life expectancy >1 year after the intervention.
* Informed consent to participate in the study after adequate information about the study before randomization and intervention.

Exclusion Criteria:

* Coronary artery disease, not suitable for both percutaneous coronary intervention (PCI) or coronary artery bypass graft surgery (CABG).
* Coronary angiogram with a SYNTAX-score >22.
* LVEF <25% without contractile reserve during dobutamine stress echocardiography.
* Porcelain aorta, which prevents open-heart surgery.
* Bicuspid valve with aorta ascendens diameter ≥45mm
* Severe femoral, iliac or aortic atherosclerosis, calcification, coarctation, aneurysm or tortuosity, which prevents transfemoral TAVR.
* Need for open heart surgery other than SAVR with or without CABG.
* Myocardial infarction within last 30 days
* Stroke or TIA within the last 30 days. NOTION-2, 01. February 2017, version 5 9
* Current endocarditis, intracardiac tumor, thrombus or vegetation.
* Ongoing severe infection requiring intravenous antibiotics.
* Unstable pre-procedural condition requiring intravenous inotropes or mechanical assist device (IABP, Impella) on the day of intervention.
* Kidney disease requiring dialysis or severely impaired lung function (FEV1 and/or diffusion capacity <40% of predicted).
* Allergy to heparin, iodid contrast agent, warfarin, aspirin or clopidogrel.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2024-02 (Actual); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Composite rate of all-cause mortality, stroke and rehospitalization (related to the procedure, the valve or heart failure) within one year after the procedure. | at one year post-procedural.
  VARC-3 definitions

SECONDARY OUTCOMES:
Procedure time | Intraoperative
  hours
Duration of index hospitalization | Number of days from admission to discharge (expected an averge of 7 days)
  days
Composite rate of all-cause mortality, stroke and rehospitalization (related to the procedure, the valve or heart failure) | at 1 month and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Composite rate of all-cause mortality, disabling stroke and rehospitalization (related to the procedure, the valve or heart failure) | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Rehospitalization both composite and individual of related to the procedure, the valve or heart failure) | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Composite rate of all-cause mortality and disabling stroke | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
All-cause mortality | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Cardiovascular mortality | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Non-cardiovascular mortality | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Stroke | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Disabling Stroke | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Non-disabling stroke | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Transient Ischemic attack | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Myocardial Infarction | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Endocarditis | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Valve Thrombosis | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Need for aortic valve re-intervention | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Bleeding (life-threatening or major) | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Vascular complication (major) | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 defintions
Acute kidney injury (stage 2 or 3) | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 defintions
Echocardiographic aortic bioprosthesis performance (degree of paravalvular leakage, valve area, mean gradient, prosthesis patient mismatch) | at discharge, 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
NYHA functional class | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  NYHA functional class
Need for permanent pacemaker | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
New onset atrial fibrillation captured on ECG | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  VARC-3 definitions
Left ventricle remodeling as assesed by echocardiography | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  Left ventricle internal diameter in diastoli
Quality of life change from baseline | at 1 and 12 months, and yearly thereafter up to 10 years post-procedure
  Kansas City Cardiomyopathy Questionnaire, scale 0 (worse) to 100 (better)

CONTACTS AND LOCATIONS:
Overall Officials: Ole De Backer, MD; PhD, Principal Investigator — Rigshospitalet, Denmark; Hans GH Thyregod, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (9):
- Denmark (2):
  - Aarhus University hospital, Aarhus
  - Rigshospitalet, Copenhagen University Hospital, Copenhagen
- Finland (3):
  - Helsinki University Central Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Turku University Hospital, Turku
- Landspital, Reykjavik, Iceland
- Haukeland University Hospital, Bergen, Norway
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jorgensen TH, Savontaus M, Willemen Y, Bleie O, Tang M, Angeras O, Niemela M, Gudmundsdottir IJ, Khokhar A, Sartipy U, Dagnegard H, Laine M, Ruck A, Piuhola J, Petursson P, Christiansen EH, Malmberg M, Olsen PS, Haaverstad R, Prendergast B, Sondergaard L, Horsted Thyregod HG, De Backer O; NOTION-2 Investigators. Three-Year Follow-Up of the NOTION-2 Trial: TAVR Versus SAVR to Treat Younger Low-Risk Patients With Tricuspid or Bicuspid Aortic Stenosis. Circulation. 2025 Nov 11;152(19):1326-1337. doi: 10.1161/CIRCULATIONAHA.125.076678. Epub 2025 Aug 30. PMID 40884768
- [Derived] Jorgensen TH, Thyregod HGH, Blankenberg S, Leon M, Sondergaard L, Prendergast B, De Backer O. The low-risk TAVR trials-A critical appraisal of the current landscape. Am Heart J. 2026 Jan;291:10-13. doi: 10.1016/j.ahj.2025.07.070. Epub 2025 Jul 29. PMID 40744194
- [Derived] Jorgensen TH, Thyregod HGH, Savontaus M, Willemen Y, Bleie O, Tang M, Niemela M, Angeras O, Gudmundsdottir IJ, Sartipy U, Dagnegaard H, Laine M, Ruck A, Piuhola J, Petursson P, Christiansen EH, Malmberg M, Olsen PS, Haaverstad R, Sondergaard L, De Backer O; NOTION-2 investigators. Transcatheter aortic valve implantation in low-risk tricuspid or bicuspid aortic stenosis: the NOTION-2 trial. Eur Heart J. 2024 Oct 5;45(37):3804-3814. doi: 10.1093/eurheartj/ehae331. PMID 38747246